CLINICAL TRIAL: NCT05941455
Title: A Prospective Multicenter Pivotal Study to Evaluate Safety and Effectiveness of Venus-Neo Surgical Aortic Valve
Acronym: METASAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jilin Venus Haoyue Medtech Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VSAF-23-02
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Aortic Valve Disease; Cardiovascular Diseases
Keywords: Heart Failure; Surgical Cardiovascular Devices
MeSH Terms: conditions — Aortic Valve Disease; Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venus-Neo group (Experimental): Procedure: surgical aortic valve replacement
  Interventions: Device: Venus-Neo Surgical Aortic Valve

INTERVENTIONS:
Device: Venus-Neo Surgical Aortic Valve — Implant of a Venus-Neo Surgical Aortic Valve

SUMMARY:
The goal of this clinical trial is to evaluate the safety, effectiveness, and performance of Venus-Neo Surgical Aortic Valve in subjects who are clinically indicated for aortic valve replacement.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-randomized interventional study to evaluate the safety, effectiveness, and performance of Venus-Neo Surgical Aortic Valve. 155 subjects are estimated to be enrolled in this study. Total enrollment period for this trial is estimated to be 1 year. Follow-up duration is estimated to be 5 years. Overall duration of the trial is estimated to be 6 years. The trial begins with the enrollment of the first subject and ends after the last subject is exited from the trial after completing the last follow-up visit at approximately 5 years, all subjects are fully monitored, all outstanding data queries are resolved.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients who are clinically indicated for aortic valve replacement
3. Patients who are willing and able to participate in the follow-up requirements, and provide written informed consent

Exclusion Criteria:

1. Previous surgical or/and transcatheter cardiac valve replacement at any site
2. Previous open-heart surgical valve repair at any site
3. Any percutaneous cardiovascular intervention (excluding diagnostic percutaneous coronary artery intervention), cardiovascular surgery, carotid surgery within 30 days
4. Untreated mitral, tricuspid, or pulmonary valve diseases requiring procedural intervention
5. Untreated clinically significant coronary artery diseases requiring revascularization
6. Acute myocardial infarct within the previous 30 days
7. Severe right heart dysfunction
8. Active infection requiring antibiotic therapy including infective endocarditis
9. Hypertrophic obstructive cardiomyopathy (HOCM)
10. Severe symptomatic carotid artery stenosis
11. Stroke or TIA within 3 months or Modified Rankin Scale ≥ 4 disability
12. Chronic kidney disease (eGFR<45 mL/min/1.73m2) or end-stage renal disease requiring chronic dialysis
13. Hematologic disorders: Leukopenia (WBC < 3000 cell/mL), anemia (Hgb < 9 g/dL), thrombocytopenia (Plt< 50,000 cell/mL), or any known blood clotting disorder, deemed clinically significant after consultation with Hematooncology specialists
14. Severe chronic lung disease
15. Previous organ transplant or currently an organ transplant candidate Anatomical
16. LVEF < 20%
17. Left ventricular end diastolic diameter (LVEDD) >70mm
18. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
19. Native aortic valve geometry and size unfavorable for study bioprosthetic valve General
20. Hemodynamics instability requiring inotropic support or intra-aortic balloon pump (IABP) or other hemodynamic support device, or any mechanical heart assistance
21. Urgent, emergency or salvage surgeries
22. Known intolerance for periprocedural/post-procedural anticoagulation or antiplatelet therapy leading to be unable to undergo index procedure per physicians' judgement
23. Life expectancy ≤ 1 year due to non-cardiac reasons
24. Planned relevant concomitant procedure within 30 days post index procedure
25. Current or recent participation (within 6 weeks prior to index procedure) in another drug or device trial
26. Pregnant, breastfeeding or intend to become pregnant within 1 year
27. Currently incarcerated or unable to give voluntary informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
primary composite safety endpoint | 1 year
  composite safety endpoint at 1 year, including: valve-related mortality, thromboembolism, aortic valve reintervention, structural valve deterioration, major paravalvular leak (defined as moderate or greater paravalvular leak or any paravalvular leak requiring intervention), valve thrombosis, endocarditis

SECONDARY OUTCOMES:
secondary composite safety endpoint | 2 through 5 Years
  safety is assessed over 1-year timeframe by comparing the occurrence of specific safety endpoints to the objective performance criteria (OPC) reported in Table I.1 in "ISO:5840-2:2021(E), Annex I, Methods of evaluating clinical data against objective performance criteria"
Occurrence of each of the following adverse events | baseline, pre-discharge, 30 days, 6 months, 12 months and annually until 5 years thereafter
  Occurrence of each of the following adverse events until 5 years, including: mortality, valve-related mortality, thromboembolism, aortic valve reintervention, structural valve deterioration, non-structural valve deterioration, all paravalvular leak, major paravalvular leak, valve thrombosis, endocarditis, all hemorrhage, major hemorrhage, bioprosthetic valve explant, hemolysis

OTHER OUTCOMES:
Clinically acceptable bioprosthetic valve performance | baseline, pre-discharge, 30 days, 6 months, 12 months and annually until 5 years thereafter
  Clinically acceptable bioprosthetic valve performance until 5 years: clinically acceptable effective orifice area (EOA), mean pressure gradient (MPG) <20mmHg, freedom from moderate or greater regurgitation (transvalvular and paravalvular), freedom from aortic valve reintervention, freedom from clinically significant bioprosthetic valve thrombosis
Procedure success | pre-discharge
  Procedure success at pre-discharge: freedom from valve-related mortality, freedom from aortic valve reintervention, intended performance of bioprosthetic valve (mean gradient <20 mmHg, peak velocity <3 m/s, and less than moderate aortic regurgitation)
New York Heart Association (NYHA) classification | baseline, pre-discharge, 30 days, 6 months, 12 months and annually until 5 years thereafter
  New York Heart Association (NYHA) classification until 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Volkmar Falk, Principal Investigator — Deutsches Herzzentrum Berlin-Charité
Locations (1):
- Deutsches Herzzentrum Berlin-Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
to publish the results